CLINICAL TRIAL: NCT06864520
Title: Valutazione Degli Effetti Benefici Di Un Prodotto Contenente Acido Γ-ammino Butirrico (GABA) Sui Disturbi Della Sindrome Climaterica CLIMATERICA
Brief Title: Evaluation of the Beneficial Effects of a Product Containing Γ-aminobutyric Acid (GABA) on Climacteric Syndrome Disorders
Acronym: GABAPAUSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Angelo Cagnacci, Full Professor Obstetric and Gynecology - Director Academic Unit of Obstetrics and Gynecology, Ospedale Policlinico San Martino
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12420
Record Dates: First submitted 2025-02-24; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Climacteric Symptoms; Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — gamma-Aminobutyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A1 with 3 capsules (Active Comparator): Tablets containing 250mg of γ-aminobutyric acid (GABA) and 50mg of Melissa extract, to be taken one at lunch and two before bedtime for 12 weeks
  Interventions: Dietary Supplement: GAMMA-AMINOBUTYRIC ACID - GABA
- Group A2 with 3 capsules (Placebo Comparator): Tablets containing microcrystalline cellulose, rice bran, bitter cocoa powder, to be taken one at lunch and two before bedtime for 12 weeks
  Interventions: Other: Placebo
- Group B1 with 2 capsules (Active Comparator): Tablets containing 250mg of γ-aminobutyric acid (GABA) and 50mg of Melissa extract, to be taken one at lunch and one before bedtime for 12 weeks
  Interventions: Dietary Supplement: GAMMA-AMINOBUTYRIC ACID - GABA
- Group B2 with 2 capsules (Placebo Comparator): Tablets containing microcrystalline cellulose, rice bran, bitter cocoa powder, to be taken one at lunch and one before bedtime for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: GAMMA-AMINOBUTYRIC ACID - GABA — Food supplement based on GABA and Melissa extract
  Arms: Group A1 with 3 capsules; Group B1 with 2 capsules
Other: Placebo — Placebo based on microcrystalline cellulose, rice bran, bitter cocoa powder
  Arms: Group A2 with 3 capsules; Group B2 with 2 capsules

SUMMARY:
The goal of this clinical trial is to learn if the food supplement based on GABA works to treat climateric symptoms. It will also learn about the safety of supplement based on GABA. The main question aims to answer:

* Does food supplement based on GABA lower the climateric symptoms, such as hot flashes, sleep, disturbances, mood swings?
* The supplement that will be administered is commonly available on the market and can be used without particular precautions. No important side effects are reported.

Researchers will compare supplement based on GABA to a placebo (a look-alike substance that contains no active ingredients) to see if supplement based on GABA works to treat climateric symptoms.

Participants will:

* Take supplement based on GABA or a placebo every day for 3 months
* Visit the clinic on day 7, 37 and 97 after enrolment for checkups and tests
* Keep a diary of number and intensity of hot flashes
* To fill scales evaluating sleep quality, anxiety, depression and quality of life

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of a commercial supplement to alleviate symptoms associated with menopause such as hot flashes, sleep disturbances, and mood swings.

Participants will be required to come to the clinic for a few visits:

* First visit in which the nature of the study will be explained, the intensity of symptoms will be assessed (using the Greene questionnaire), and the inclusion and exclusion criteria for participation in the study will be assessed. If the participant is eligible for the study, they will be asked to fill out a diary for the next 7 days in which to indicate the daily number and intensity of hot flashes;
* Second visit in which the hot flash diary will be collected and the following questionnaires will be submitted: Greene Scale to determine climacteric symptoms; STAI-Y1 to determine state anxiety (20 questions); SDS to determine the presence of depression (20 questions); PSQI to determine the quality of sleep (9 questions); MenQoL, Quality of life (29 questions). At this visit, a new diary will be provided, in which the number and intensity of hot flashes during the last 7 days before the next visit must be reported, and the product to be taken for the following month will be provided; neither the participant nor the investigator are aware of the product provided: study product or placebo;
* Third visit, in which the hot flash diary and the product package delivered at the previous visit will be collected. The participant will have to fill in all the questionnaires completed at the previous visit and will also be asked about the degree of satisfaction with the first 30 days of treatment. At this visit, a new diary will be provided, in which the number and intensity of hot flashes during the last 7 days before the next visit must be reported, and the product to be taken for the following two months will be provided;
* Fourth visit, in which the hot flash diary and the product package delivered at the previous visit will be collected. The participant will have to fill out all the questionnaires completed at the previous visit and will also be asked about the degree of satisfaction with the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Physiological or iatrogenic menopause (amenorrhea for at least 12 months or for 6 months with FSH ≥40 IU/L)
* Greene Index value ≥ 15

Exclusion Criteria:

* Patients who do not consent to the study
* Patients who have used hormone replacement therapy in the last 3 months
* Patients who have used phytotherapeutics in the last 3 months
* Patients who have used acupuncture in the last 3 months
* Uncompensated hyper or hypothyroidism
* Acute phase of endocrine pathologies
* Patients with major psychiatric disorders
* Addiction to opioids or alcohol
* Glaucoma
* Active liver disease
* Use of antidepressants, benzodiazepines or any neuroactive drug
* Known allergy to the components of the treatment being studied

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of the Greene Climacteric Scale Score | From enrollment to the end of treatment at 12 weeks
  The Greene Scale is a verified measurement tool which provides a brief measure of menopause symptoms. It is composed of 21 items evaluating the bother of climacteric symptoms with a score for each symptom from none (value of 0) to mild (value of 1) to moderate (value of 2) to intense (value of 3). The total score of the ranges from 0 to 63, higher values corresponding to more intense climacteric symptoms. A value equal or greater than 15 indicates the presence of climacteric symptoms

SECONDARY OUTCOMES:
Assessment of anxiety with the State-Trait Anxiety Inventory-Y1 (STAI-Y1) questionnaire | From enrollment to the end of treatment at 12 weeks
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of state (Y1) of anxiety with 20 items. It can be used to diagnose anxiety and to distinguish it from depressive syndromes. All items are rated on a 4-point scale (with 1 = not at all and 4 = very much) and the total score is between 20 and 80 with a threshold value predictive of anxious symptoms set at 40. Higher scores are positively correlated with higher levels of anxiety
Assessment of sleep quality with the Pittsburgh Sleep Quality Index (PSQI) questionnaire | From enrollment to the end of treatment at 12 weeks
  The Pittsburgh Sleep Quality Index assesses sleep quality and disturbances. The global score ranges between 0 and 21, where higher scores indicate worse sleep quality
Reduction in the number and intensity of hot flashes, assessed with a daily diary 7 days before follow up | From enrollment to the end of treatment at 12 weeks
  Participants report in their daily diary the number and intensity of hot flashes, rating them on a 3-point scale (1 = mild, 2 = moderate, and 3 = severe).
Assessment of quality of life with the Menopause-specific Quality of Life (MenQoL) questionnaire | From enrollment to the end of treatment at 12 weeks
  The MENQOL consists of a total of 29 items in a Likert-scale format. Each item assesses the impact of one of four domains of menopausal symptoms: vasomotor, psychosocial, physical, and sexual. Items pertaining to a specific symptom are rated as present or not present, and if present, how bothersome on a zero (not bothersome) to six (extremely bothersome) scale. The possible score on any item ranges from one to eight, where higher score indicates higher symptoms
Comparison of the efficacy of two dosages | From enrollment to the end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Cagnacci, MD, PhD, Principal Investigator — Clinica Ostetrica e Ginecologica, IRCCS-Ospedale San Martino di Genova
Locations (1):
- Ospedale San Martino, Genova, Italia, Italy